CLINICAL TRIAL: NCT00083772
Title: The Use of Nesiritide in the Management of Acute Diastolic Heart Failure
Brief Title: Use of Nesiritide in the Management of Acute Diastolic Heart Failure
Status: Terminated | Phase: Phase 4 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2003-0782
Record Dates: First submitted 2004-06-02; First posted 2004-06-03 (Estimated); Last update posted 2018-11-07 (Actual); Status verified 2018-11

CONDITIONS: Heart Failure; Cardiovascular Disease; Acute Heart Failure; Diastolic Heart Failure; Congestive Heart Failure; Heart Disease
Keywords: Heart failure; Diastolic heart failure; Congestive heart failure; Nesiritide; Natrecor; Left ventricular (LV) diastolic function; Fatigue; Shortness of breath; Edema; Heart disease
MeSH Terms: conditions — Heart Failure; Cardiovascular Diseases; Heart Failure, Diastolic; Heart Diseases; Fatigue; Dyspnea; Edema | interventions — Natriuretic Peptide, Brain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): Nesiritide
  Interventions: Drug: Nesiritide

INTERVENTIONS:
Drug: Nesiritide — Initial dose by vein of 2 mcg/kg then infusion by vein of 0.01 mcg/kg/min continuously for 48 hours.
  Other Names: Natrecor

SUMMARY:
Primary objective is to assess the effect of nesiritide in decreasing left ventricular (LV) filling pressure, defined as pulmonary artery capillary wedge pressure (PCWP) in a group of patients admitted with acute diastolic heart failure.

Secondary objectives include: improvement in symptoms, exercise tolerance, improvement in Doppler diastolic filling parameters in patients with diastolic heart failure.

DETAILED DESCRIPTION:
Patients with diastolic heart failure often have high pressure in their heart and lungs and many symptoms such as shortness of breath, low energy, fluid retention, and fatigue. Decreasing the pressure in the heart and lungs may help these patients feel better. The drug nesiritide was designed to help treat heart failure. It has also been shown to help decrease the pressure in the lungs.

Before treatment starts, you will be asked questions about your medical history and about any medications you are currently taking. You will have a complete physical exam. You will have an electrocardiogram (ECG - a test that measures the electrical activity of the heart) and routine blood tests (about 2 teaspoons). You will have an ultrasound on your heart called an echocardiogram to measure your heart function and the pressures in your lungs. Your ability to breathe will be evaluated. With the aid of the research nurse, you will have a 6-minute walk test. You may stop or sit down at any time during the test. This test is being done to evaluate your energy level. You will also be asked to complete a questionnaire about your symptoms. This questionnaire should take no more than 10 minutes to complete.

In order to measure the pressure in your heart and lungs, you will have a procedure called a "right heart catheterization". This is a procedure that may have been done as part of your standard of care even if you were not enrolled in this study. For this procedure, a small tube will be placed in a vein in your neck. A longer tube will be inserted into the first tube and fed through the vein and into your heart. This tube will be used to measure the pressure in your heart and lungs. After the pressures are measured, you will receive treatment with nesiritide during the right heart catheterization procedure.

Nesiritide will be given as a continuous infusion (for 48 hours) by vein. The pressures in your heart and lungs will be measured again at 15, 30, then 60 minutes after you begin to receive nesiritide. The tubes will then be removed from your heart. You will be awake during this procedure and lying flat on your back. An anesthetic will be used to numb the area of your neck where the tube is placed. The entire procedure (including treatment) should take no longer than 1 hour. You will have an ultrasound of your heart performed immediately before and after the right heart catheterization.

Within 15 minutes of the end of the procedure the echocardiogram, the 6-minute walk test, and the questionnaire about your symptoms will be repeated and your breathing will be re-evaluated.

The nesiritide infusion will remain going through a vein in your arm for the next 48 hours. During this infusion you will remain in the hospital on telemetry floor so that researchers can monitor your blood pressure and watch for irregular heartbeat. After you have received this drug for 48 hours, the drug will be stopped. Within 24 hours after stopping treatment, an echocardiogram and a 6-minute walk test will be performed. You will also answer questions about your breathing and your quality of life. These should take no more than 15 minutes of your time to complete.

You will be taken off study if your condition gets worse or intolerable side effects occur.

At 2 and 4 weeks after your hospitalization and the right heart procedure, you will have follow-up visits scheduled. At these visits, you will have a complete physical exam, and possibly have blood work done if required by the doctor as part of your routine care. A blood test to check a BNP (B-type natriuretic peptide) level will also be performed . This is a special blood test to give researchers information about your heart and how much extra fluid you may be carrying with you because of your heart disease. Only 1 teaspoon of blood is needed for this test although up to 3 teaspoons of blood may need to be drawn depending of what blood tests your doctor orders at the follow-up visits.

This is an investigational study. Nesiritide is FDA approved and is commercially available for the treatment of heart failure. However, the use of nesiritide for diastolic heart failure is under research. About 20 patients will take part in this study. All will be enrolled at UTMDACC.

ELIGIBILITY:
The patient population recruited for this study will include patients being admitted for acute congestive heart failure. Eligible patients include those who have near normal LV systolic function.

Inclusion Criteria:

* Age 18 to 85 years old
* Admitted with acute heart failure determined by: symptoms of fatigue; shortness of breath; edema; physical evidence of volume overload; and/or pulmonary edema by CXR
* LVEF > or = 40% on recent (< or = 1 month) echo or MUGA
* NYHA class III or IV on admission
* Baseline systolic blood pressure > 90 mm Hg
* Baseline BNP level > 100 pg/ml
* Able to sign informed consent and return for follow-up assessments

Exclusion Criteria:

* Patients with clinically significant hypotension (defined as a systolic blood pressure (SBP) <90 mm Hg)
* Active infection/sepsis as defined by fever > 101.5 F, currently on IV antibiotics
* Creatinine greater than 3.0 mg/dl
* LV ejection fraction < 40% (must be done within the last 30 days prior to signing consent)
* Significant valvular disease or constrictive cardiomyopathy
* Severe Thrombocytopenia (as defined by platelets less than 20,000) or INR > 1.6
* Hypersensitivity to nesiritide or any of its components.
* Pulmonary capillary wedge pressure (PCWP) <16 mmHg
* If patient is of child-bearing age, a pregnancy test will be performed, and the patient is excluded if pregnancy test is positive.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2004-05-17 (Actual); Primary Completion 2006-04-24 (Actual); Study Completion 2006-04-24 (Actual)

PRIMARY OUTCOMES:
Effectiveness of nesiritide in improving symptoms, including pressure in heart and lungs, related to diastolic heart failure (condition where heart muscle is stiff and not able to relax completely, causing the pressures in heart to increase). | 2 Years

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Bernard Durand, MD, Study Chair — UT MD Anderson Cancer Center

REFERENCES:
- [Background] Krishnaswamy P, Lubien E, Clopton P, Koon J, Kazanegra R, Wanner E, Gardetto N, Garcia A, DeMaria A, Maisel AS. Utility of B-natriuretic peptide levels in identifying patients with left ventricular systolic or diastolic dysfunction. Am J Med. 2001 Sep;111(4):274-9. doi: 10.1016/s0002-9343(01)00841-5. PMID 11566457
- [Background] Cheng V, Kazanagra R, Garcia A, Lenert L, Krishnaswamy P, Gardetto N, Clopton P, Maisel A. A rapid bedside test for B-type peptide predicts treatment outcomes in patients admitted for decompensated heart failure: a pilot study. J Am Coll Cardiol. 2001 Feb;37(2):386-91. doi: 10.1016/s0735-1097(00)01157-8. PMID 11216951
- [Background] Zile MR, Gaasch WH, Carroll JD, Feldman MD, Aurigemma GP, Schaer GL, Ghali JK, Liebson PR. Heart failure with a normal ejection fraction: is measurement of diastolic function necessary to make the diagnosis of diastolic heart failure? Circulation. 2001 Aug 14;104(7):779-82. doi: 10.1161/hc3201.094226. PMID 11502702
- [Background] Mills RM, Hobbs RE, Young JB. "BNP" for heart failure: role of nesiritide in cardiovascular therapeutics. Congest Heart Fail. 2002 Sep-Oct;8(5):270-3. doi: 10.1111/j.1527-5299.2002.01154.x. PMID 12368590
- [Background] Publication Committee for the VMAC Investigators (Vasodilatation in the Management of Acute CHF). Intravenous nesiritide vs nitroglycerin for treatment of decompensated congestive heart failure: a randomized controlled trial. JAMA. 2002 Mar 27;287(12):1531-40. doi: 10.1001/jama.287.12.1531. PMID 11911755
- See also: MD Anderson Cancer Center, Department of Cardiology — http://www.mdanderson.org/departments/cardiology/